CLINICAL TRIAL: NCT05795881
Title: Effect of Continuous Versus Cyclic Daytime Enteral Nutrition on Circadian Rhythms in Critical Illness: CIRCLES Study
Brief Title: Effect of Continuous Versus Cyclic Daytime Enteral Nutrition on Circadian Rhythms in Critical Illness
Acronym: CIRCLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, David van westerloo, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P22.080
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Intensive Care Unit; Circadian Rhythm; Sleep; Enteral Nutrition
Keywords: Randomized Controlled Trial
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Investigator-Initiated Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): continuous enteral nutrition: 24 hours a day (standard of care)
- Intervention group (Experimental): cyclic daytime enteral nutrition: between 8 a.m. and 8 p.m. (same amount of nutrition as control group)
  Interventions: Other: Cyclic daytime enteral nutrition

INTERVENTIONS:
Other: Cyclic daytime enteral nutrition — The allocated feeding schedule is followed from the start of enteral nutrition after ICU admission until discharge from the ICU.
  Arms: Intervention group

SUMMARY:
Disruption of circadian rhythms is frequently observed in patients in the intensive care unit (ICU) and is associated with worse clinical outcomes. The ICU environment presents weak and conflicting timing cues to the circadian clock, including continuous enteral nutrition. The goal of this clinical trial is to evaluate the effect of timing of enteral nutrition on the circadian rhythm in critically ill patients. Patients admitted to the intensive care unit will be allocated to receive either continuous or cyclic daytime (8am to 8 pm) enteral feeding. Differences in circadian rhythms will be assessed by 24h patterns in core body temperature, heart rate variability, melatonin and peripheral clock gene expression. Secondary outcomes include depth of sleep, glucose variability and incidence of feeding intolerance. This study is expected to contribute to the optimalisation of circadian rhythms in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Receiving of or intention to start enteral nutrition via nasogastric or nasoduodenal tube
* Arterial line
* Expected duration of ICU admission > 48 hours

Exclusion Criteria:

* Receiving parenteral nutrition
* Prior night-time (20.00h - 8.00h) enteral tube feeding within the same hospitalization before study inclusion
* Readmission to ICU with prior study inclusion
* Chronic enteral tube feeding prior to current admission
* Presence of one or more contraindications of enteral feeding and/or at significant risk for gastrointestinal tolerance according to standard protocol (including but not limited to gastrointestinal haemorrhage, intestinal ischemia or necrosis, impaired digestive tract integrity due to obstruction or perforation, gastrectomy, enterectomy, history of gastroparesis or oesophageal dysmotility or expected surgery within 24 hours)
* Patients with glycaemic emergency (including but not limited to hyperglycaemic hyperosmolar nonketotic coma, diabetic ketoacidosis, severe hypoglycaemia resulting in ICU admission) or patients controlling their glucose levels and insulin dosing via continuous glucose monitoring
* Expected death within 24 hours
* Do-not-resuscitate (DNR) order
* Treatment with extracorporeal membrane oxygenation
* Severe neurological damage (significant neurological abnormalities such as bleeding, ischemia, neurotrauma or severe encephalopathy with Glasgow Coma Scale ≤ 8)
* Suspected or confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Amplitude of 24-h rhythm of core body temperature | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Acrophase 24-h rhythm of core body temperature | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis

SECONDARY OUTCOMES:
Amplitude of 24-h rhythm of plasma melatonin levels | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Acrophase of 24-h rhythm of plasma melatonin levels | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Amplitude of 24-h rhythm in heart rate variability | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Acrophase of 24-h rhythm in heart rate variability | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Amplitude of 24-h rhythm in systolic blood pressure | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Acrophase of 24-h rhythm in systolic blood pressure | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Amplitude of 24-h rhythm in heart rate | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Acrophase of 24-h rhythm in heart rate | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Determined by cosinor analysis
Peripheral clock gene expression | Day 3 (12 p.m.) to day 4 (12 a.m.) after start of the study intervention (= start of enteral nutrition)
  Time of day-dependent difference in clock gene expression in PBMCs isolated from blood samples collected at 12 p.m. and 12 a.m.
Depth of sleep | Day 3 (8 a.m.) to day 4 (8 a.m.) after start of the study intervention (= start of enteral nutrition)
  Daytime (8 a.m. to 8 p.m.) to nighttime (8 p.m. to 8 a.m.) ratio of gamma to delta spectral power ratio in EEG measured with a sleep headband
Mean daily rate of hyperglycaemia/hypoglycaemia | From start of study intervention (enteral nutrition) to end of study intervention
  Hypoglycaemia is defined as glucose levels < 3.5 mmol/L, hyperglycaemia is defined as glucose levels >10 mmol/L
Mean daily glucose variability | From start of study intervention (enteral nutrition) to end of study intervention
  Mean of standard deviation of glucose levels per day
Mean daily insulin administration | From start of study intervention (enteral nutrition) to end of study intervention
  Mean of number of insulin units used per day
Mean daily caloric intake | From start of study intervention (enteral nutrition) to end of study intervention
  Mean of percentage of recommended calories that patient receives per day of interest during study period
Daily rates of gastric retention | From start of study intervention (enteral nutrition) to end of study intervention
  Gastric retention is defined as gastric residual volume > 200 mL
28-day mortality | Up to 28 days
  28-day mortality
Days on mechanical ventilation | From ICU admission to ICU discharge
  Days on mechanical ventilation
ICU length of stay | From ICU admission to ICU discharge
  ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: David J van Westerloo, PhD, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Immediately following publication, the individual participant data that underlie the results reported in the published article will be shared after deidentificiation. The data will be shared upon request with researchers who wish to access the data for any purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available immediately following publication.
Access Criteria: to be announced

REFERENCES:
- [Background] Kouw IWK, Heilbronn LK, van Zanten ARH. Intermittent feeding and circadian rhythm in critical illness. Curr Opin Crit Care. 2022 Aug 1;28(4):381-388. doi: 10.1097/MCC.0000000000000960. Epub 2022 Jul 5. PMID 35797531
- [Derived] Hiemstra FW, van Gent MF, de Jonge E, van Westerloo DJ, Kervezee L. Effect of cyclic daytime versus continuous enteral nutrition on circadian rhythms in critical illness (CIRCLES): Study protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Jul;154:107927. doi: 10.1016/j.cct.2025.107927. Epub 2025 Apr 27. PMID 40300711